CLINICAL TRIAL: NCT04023305
Title: Sevoflurane pharmacokInetics During Inhaled Sedation Relies on the Morphotype of ARDS in ICU Patients
Brief Title: Sevoflurane PharmacokInetics in ARDS
Acronym: SPIDERMAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPIDERMAN Study; 2018-003511-21 (EudraCT Number)
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Nonfocal Acute respiratory distress syndrome; Focal Acute respiratory distress syndrome; Sevoflurane; Pharmacokinetics; Mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Inhaled sedation with sevoflurane, will be vaporized via the miniaturized Anesthesia Conserving Device (AnaConDa-S®, Sedana Medical, Uppsala, Sweden).
  Sevoflurane infusion rate will be adapted from manufacturer's instructions in order to reach a target of expired sevoflurane fraction (FEsevo) of 0.8-1.1.
  Mechanical ventilation will be protocolized in both arms, based on recent results of a RCT from our group, in which 90-day survival was improved in patients with nonfocal ARDS when an individualized ventilation strategy was applied, compared to the ARDSNet strategy (PEEP set according to FiO2). We will recommend sites wait at least 12 hours before proning, as in the PROSEVA study.
  In both groups, patients will receive cisatracurium besylate for neuromuscular blockade, and deep sedation will be protocolized to Richmond Agitation-Sedation Scale (RASS) of -4 to -5 (Ramsay of 5-6, or Riker of 1-2) before starting, and during, the cisatracurium besylate infusion.
Who Masked: Outcomes Assessor
Masking Description: It is an open label trial because the patients are included from a group depending to the morphotype of ARDS. However, all subsequent evaluations will be conducted by clinical research staff according to the attributed group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonfocal ARDS (Experimental): ARDS patient with nonfocal lung imaging phenotype
  Interventions: Drug: Deep sedation by Sevoflurane on the Morphotype of ARDS in ICU patieNts
- Focal ARDS (Experimental): ARDS patient with focal lung imaging phenotype
  Interventions: Drug: Deep sedation by Sevoflurane on the Morphotype of ARDS in ICU patieNts

INTERVENTIONS:
Drug: Deep sedation by Sevoflurane on the Morphotype of ARDS in ICU patieNts — Pharmacokinetic of inhaled sevoflurane used for sedation

SUMMARY:
The main objective of this study is to compare the pharmacokinetic models of sevoflurane-induced sedation during ARDS depending on the lung imaging phenotype (focal vs nonfocal phenotypes) The authors hypothesized that sevoflurane used for inhaled sedation could have distinct pharmacokinetic profiles depending on lung imaging phenotypes (focal vs nonfocal) during ARDS in ICU patients.

DETAILED DESCRIPTION:
Adult patients admitted to the ICU within 12 hours of moderate-severe ARDS onset and under sedation with sevoflurane will be enrolled in the study with inclusion criteria. They will be enrolled, depending on their morphotype (focal or nonfocal), as routinely assessed in participating centers using CT-scan, chest x-ray and/or lung ultrasound.

These patients will receive inhaled sevoflurane as a standard practice of sedation that is routinely used in participating ICUs. After inclusion, the mechanical ventilation protocol must be initiated within two hours (if not already being used). In both groups, deep sedation followed by neuromuscular blockade must be initiated within four hours of inclusion.

Adult patients admitted to the ICU within 12 hours of moderate-severe ARDS onset and under sedation with sevoflurane will be enrolled in the study with inclusion criteria. They will be enrolled, depending on their morphotype (focal or nonfocal), as routinely assessed in participating centers using CT-scan, chest x-ray and/or lung ultrasound.

These patients will receive inhaled sevoflurane as a standard practice of sedation that is routinely used in participating ICUs. After inclusion, the mechanical ventilation protocol must be initiated within two hours (if not already being used). In both groups, deep sedation followed by neuromuscular blockade must be initiated within four hours of inclusion.

Blood sample will be collected at different times after the onset of sevoflurane administration and after its cessation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence for ≤ 12 hours of all of the following conditions, within one week of a clinical insult or new or worsening respiratory symptoms :

a PaO2/FiO2 < 200 mmHg with positive end-expiratory pressure (PEEP) ≥ 8 cmH2O (or, if arterial blood gas not available : SpO2/FiO2 ratio that is equivalent to a PaO2/FiO2 < 200 mmHg with PEEP ≥8 cmH2O, and a confirmatory SpO2/FiO2 ratio between 1-6 hours after the initial SpO2/FiO2 ratio determination) b Bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules c Respiratory failure not fully explained by cardiac failure or fluid overload; need objective assessment (e.g., echocardiography) to exclude hydrostatic edema if no risk factor present

Exclusion Criteria:

* Lack of informed consent
* Continuous sedation with inhaled sevoflurane at enrollment
* Currently receiving ECMO therapy
* Chronic respiratory failure defined as PaCO2 > 60 mmHg in the outpatient setting
* Home mechanical ventilation (non-invasive ventilation or via tracheotomy) except for CPAP/BIPAP used solely for sleep-disordered breathing
* Body mass index > 40 kg/m2
* Chronic liver disease defined as a Child-Pugh score of 12-15
* Expected duration of mechanical ventilation < 48 hours
* Tidal volume of 6 mL/kg predicted body weight (PBW) below 200 mL
* Decision to withhold life-sustaining treatment; except in those patients committed to full support except cardiopulmonary resuscitation
* Moribund patient, i.e. not expected to survive 24 hours despite intensive care
* Burns > 70% total body surface
* Previous hypersensitivity or anaphylactic reaction to sevoflurane
* Medical history of malignant hyperthermia
* Suspected or proven intracranial hypertension
* Know pregnancy - Pregnancy testing will be systematically performed to rule out pregnancy in female patients of reproductive age
* Enrollment in another interventional ARDS trial with direct impact on sedation and PEEP
* Endotracheal ventilation for greater than 120 hours (5 days)
* PaO2/FiO2 (if available) > 200 mmHg after meeting inclusion criteria and before start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of sevoflurane | 5 minutes after the detection by the monitor of sevoflurane (0.1%) in the breathing circuit
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 30 minutes after the detection by the monitor of sevoflurane (0.1%) in the breathing circuit
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 1 hour after the detection by the monitor of sevoflurane (0.1%) in the breathing circuit
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 6 hours after the detection by the monitor of sevoflurane (0.1%) in the breathing circuit
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 24 hours after the detection by the monitor of sevoflurane (0.1%) in the breathing circuit
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 48 hours after the detection by the monitor of sevoflurane (0.1%) in the breathing circuit
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 5 minutes after the cessation of sevoflurane administration
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 30 minutes after the cessation of sevoflurane administration
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 1 hour after the cessation of sevoflurane administration
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 4 hours after the cessation of sevoflurane administration
  Plasma concentrations of sevoflurane
Plasma concentrations of sevoflurane | 6 hours after the cessation of sevoflurane administration
  Plasma concentrations of sevoflurane

SECONDARY OUTCOMES:
Plasma concentration of hexafluoroisopropanolol | Until sedation can be definitely interrupted or until day 7
  Plasma concentration of hexafluoroisopropanolol
Fraction of inspired sevoflurane | Until sedation can be definitely interrupted or until day 7
  Fraction of inspired sevoflurane
Fraction of expired sevoflurane | Until sedation can be definitely interrupted or until day 7
  Fraction of expired sevoflurane
Dose of sevoflurane | Until sedation can be definitely interrupted or until day 7
  Dose of sevoflurane (mg/l)
Infusion duration of sevoflurane | Until sedation can be definitely interrupted or until day 7
  Infusion duration of sevoflurane (min)
Infusion rate of remifentanil | Until sedation can be definitely interrupted or until day 7
  Infusion rate of remifentanil
Values of a bispectral index | Until sedation can be definitely interrupted or until day 7
  Values of a bispectral index

CONTACTS AND LOCATIONS:
Overall Officials: Raiko Blondonnet, MD, MSc, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (3):
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU, Clermont-Ferrand
  - APHP - University hospital of Saint-Louis, Paris